CLINICAL TRIAL: NCT00829803
Title: A Prospective Randomized Double Blinded Study Assessing Indices of SNAP vs VISTA on Surgical Patients Undergoing General Anesthesia
Brief Title: A Study to Assess Indices of SNAP vs VISTA on Surgical Patients Undergoing General Anesthesia
Acronym: Precision GA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SIS-SNAP-2008-01US
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2011-06

CONDITIONS: Anesthesia, General
Keywords: To acquire developmental data to prospectively support SNAP; II index ranges at the studied anesthetic states.
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- SNAP Monitor EEG signals (Experimental)
  Interventions: Device: SNAP monitor; Bispectral Index Monitor (BIS Monitor)
- BIS Monitor EEG signals (VISTA) (Active Comparator)
  Interventions: Device: SNAP monitor; Bispectral Index Monitor (BIS Monitor)

INTERVENTIONS:
Device: SNAP monitor; Bispectral Index Monitor (BIS Monitor) — Intended to monitor the state of the brain by data acquisition of EEG signals.
  Other Names: SNAP II monitor; BIS Monitor

SUMMARY:
Establish the range of index values for the SNAP II corresponding to each anesthetic state studied.

DETAILED DESCRIPTION:
Index values for the SNAP II monitor will be identified with each corresponding anesthetic state studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery requiring general anesthesia
* Open or laparoscopic procedures
* Cases anticipated to be less than 4 hours in duration
* In-patient and out-patient subjects
* Patients and cases manageable with LMA. Cases manageable with ET tube are also allowed with the condition that only a minimal dose of short-acting NMBA is used at intubation and not throughout the case.
* Local analgesia at incision site is permitted.
* Males and Females between 18 and 65 years of age, inclusive.
* BMI<40 and body mass>41 kg
* Patients who have signed the informed consent.
* Able to receive Informed Consent through subjects native language providing that a native language speaker delivers the Informed Consent.
* ASA Stratification I - III

Exclusion Criteria:

* Any subject failing to fulfill all inclusion criteria
* ASA stratification >= IV
* Subject is a prisoner.
* Patients presenting with evidence of recent trauma, active infection, neurological disorder, seizure disorder, dementia or have been diagnosed with Alzheimer's disease
* Subjects with cardiac or gastric pace makers
* Pregnant women as identified by institutional SOP for female of child-bearing age
* Patients that will not sign an informed consent form
* Patients with previous adverse incidents with anesthesia, including awareness
* Patients undergoing surgery on the head or neck
* Subjects currently taking psychoactive medications as part of routine medical care within the past 7 days
* Subjects that require and/or receive any of the psychotherapeutic agents or psychotropic drugs below, in the treatment of mental illness, and have taken such treatment within the past 7 days.
* Benzodiazepines
* MAOI inhibitors
* Selective serotonin reuptake inhibitors (SSRIs)
* Tricyclic antidepressants
* Lithium
* Neuroleptic agents
* Central nervous system stimulants.
* Subjects with a known history of alcohol or narcotic abuse within 6 months prior to screening OR subjects reporting narcotic or narcotic medication use with 24 hours prior to surgery.
* Subjects requiring neurophysiologic monitoring
* Subjects requiring TIVA
* Subjects requiring prolonged use of NMBA beyond dose required for intubation
* Subjects requiring ketamine
* Subjects receiving spinal, epidural, or other nerve blocks
* Subjects having any condition or severe illness that to the Principal Investigator's discretion would interfere with study assessments OR other severe acute or chronic medical or psychiatric condition that may interfere with the interpretation of study results and, in the judgment of the investigator, and would make the subject inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
SNAP Index values corresponding to anesthetic states: Pre-induction (baseline), loss of response, anesthesia maintenance, first purposeful response after anesthesia is discontinued, at extubation or LMA removal | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Bergese, M.D., Study Chair — Ohio State University
Locations (4):
- United States (4):
  - University Of Miami, Miami, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Beaumont Hospital, Royal Oak, Michigan
  - The Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Bergese SD, Uribe AA, Puente EG, Marcus RL, Krohn RJ, Docsa S, Soto RG, Candiotti KA. A Prospective, Multicenter, Single-Blind Study Assessing Indices of SNAP II Versus BIS VISTA on Surgical Patients Undergoing General Anesthesia. JMIR Res Protoc. 2017 Feb 3;6(2):e15. doi: 10.2196/resprot.6741. PMID 28159731